CLINICAL TRIAL: NCT01574001
Title: Comparison of Smoking Cessation Interventions of Different Intensities in Patients With First Ever Ischemic Stroke.
Brief Title: Smoking Cessation Interventions in Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Psychiatry and Neurology, Warsaw (Other)
Responsible Party: Principal Investigator, Halina Sienkiewicz-Jarosz, Principal Investigator, Institute of Psychiatry and Neurology, Warsaw
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IPIN-01; UMO-2011/01/B/NZ7/05402 (Other Grant/Funding Number: National Science Center, Poland)
Record Dates: First submitted 2012-04-01; First posted 2012-04-10 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2012-04

CONDITIONS: Ischemic Stroke
Keywords: ischemic stroke; smoking cessation; antismoking interventions
MeSH Terms: conditions — Ischemic Stroke; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Antismoking intervention with minimal early follow-up (Experimental): an intervention according to the "5A's" model with one follow-up visit within one week after discharge from the hospital; follow-up assessment will include two visits: 3 and 12 months after stroke
  Interventions: Behavioral: Antismoking intervention with minimal early follow-up
- Antismoking intervention with no early follow-up (Active Comparator): an anti-smoking intervention in line with the "5A's" method without early follow-up; follow-up assessment will be limited to two visits: 3 and 12 months after stroke
  Interventions: Behavioral: Antismoking intervention with no early follow-up
- Antismoking intervention with intensive early follow-up (Experimental): an anti-smoking intervention in line with the "5A's" method will be given, including four follow-up visits within 6 weeks after discharge from the hospital (week 1, week 2, week 4, week 6 after stroke); follow-up assessment will include two visits: 3 and 12 months after stroke
  Interventions: Behavioral: Antismoking intervention with intensive early follow-up

INTERVENTIONS:
Behavioral: Antismoking intervention with no early follow-up — an anti-smoking intervention in line with the "5A's" method without early follow-up; follow-up assessment will be limited to two visits: 3 and 12 months after stroke
  Arms: Antismoking intervention with no early follow-up
Behavioral: Antismoking intervention with minimal early follow-up — Anti-smoking intervention in line with the "5A's" method (Ask, Advice, Assess, Assist, Arrange follow-up. The intervention will be carried out 5-7 days after stroke, before the planned discharge from the hospital. Seven days after discharge from a stroke unit a brief telephone/personal advice will be given aimed to motivate patients to quit smoking; follow-up assessment will include two visits: 3 and 12 months after stroke
  Arms: Antismoking intervention with minimal early follow-up
Behavioral: Antismoking intervention with intensive early follow-up — an anti-smoking intervention in line with the "5A's" method will be given, including four follow-up visits within 6 weeks after discharge from the hospital (week 1, week 2, week 4, week 6 after stroke); follow-up assessment will include two visits: 3 and 12 months after stroke
  Arms: Antismoking intervention with intensive early follow-up

SUMMARY:
The primary objective of the present randomized controlled trial is to compare the effectiveness of three anti-smoking interventions of different intensities. It has been hypothesised that early follow-up visits facilitate post-stroke smoking cessation in patients hospitalized because of first-ever ischemic stroke.

DETAILED DESCRIPTION:
BACKGROUND: It is well known, that continued smoking after stroke increases the risk of death and stroke recurrence within a few years after the first stroke. Searching for more efficient methods of antismoking interventions is therefore justified.

OBJECTIVES: The primary objective of the present study is to compare the effectiveness of three anti-smoking interventions of different intensities.

DESIGN: Randomized, controlled trial.

METHODS: Study participants will be recruited among patients of neurological clinics of Institute of Psychiatry and Neurology, hospitalized because of their first in a lifetime ischemic stroke. All stroke patients will be screened regarding their smoking status. The subjects will be patients smoking cigarettes immediately before their first-ever stroke, able to understand the research protocol procedures and able to cooperate during the investigation.

Antismoking interventions will be based on the "5A's" method. Study participants will be randomized to one of three interventions differing in follow-up intensity.

ELIGIBILITY:
Inclusion Criteria:

* Patients smoking immediately prior to stroke
* The first in the lifetime ischemic stroke
* Ability to understand the research protocol procedures and cooperation during the investigation
* Reported availability of and declaration to participate in follow-up
* Informed consent to participate in the study

Exclusion Criteria:

* Severe stroke
* Stroke onset more than 3 weeks before admission
* History of previous stroke with clinical symptoms
* Hemorrhagic stroke
* Diagnosis of dementia or presence of other neurological disease (Parkinson's disease, amyotrophic lateral sclerosis, multiple sclerosis, Huntington's chorea, a previous subarachnoid haemorrhage, meningitis, cerebral trauma in an interview)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Smoking cessation rate | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Halina Sienkiewicz-Jarosz, M.D., PhD, Principal Investigator — 1st Department of Neurology, Institute of Psychiatry and Neurology, 9 Sobieskiego Str., 02-957 Warsaw, Poland
Locations (1):
- Institute of Psychiatry and Neurology, Warsaw, Poland